CLINICAL TRIAL: NCT01529320
Title: Pilot, Phase I, Single Blind Trial to Assess Itch Behavior in Nickel Sulphate Sensitized Volunteers. (PRURITUS- Nimpa Study).
Brief Title: Assess Itch Behavior in Nickel Sulphate Sensitized Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion IMIM (Other)
Collaborators: Adknoma Health Research (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Ana Maria Gimenez Arnau, MD, Fundacion IMIM
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: GIM-MPA-2011-01; 2011-005284-25 (EudraCT Number)
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Allergic Contact Eczema
MeSH Terms: interventions — methylprednisolone aceponate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adventan® (metilprednisolona aceponato 0,1%) (Experimental)
  Interventions: Drug: Adventan® (methylprednisolone aceponate 0,1%)

INTERVENTIONS:
Drug: Adventan® (methylprednisolone aceponate 0,1%) — Doses: 1/4 FTU (Finger Tip Unit) during 5 days (Day 7-Day 11). Procedure: Patch Test (Nickel sulphate 5%) during 2 days (Day 0- Day 2.

SUMMARY:
Determine the mean time to itch relief from the start of treatment with topic methylprednisolone aceponate.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years old.
2. Subjects with a history of diagnosis of sensitization to Nickel sulphate.
3. Delayed type hypersensitivity demonstrated by positive reaction with epicutaneous or patch test.
4. Skin Phototype II-III.
5. Women with fertile age and a negative result in the pregnancy test before inclusion. Women must use an adequate contraceptive method during the study.
6. Written informed consent prior to inclusion.
7. Able and willing to comply with protocol procedures and to follow the investigator's instructions.

Criteria for treatment initiation: At day 7, before starting treatment, subjects must meet the inclusion criteria and all the following criteria: ≥ 3 VAS and eczema intensity of (+ +) or (+++) according to ICDRG scale.

Exclusion Criteria:

1. Active cutaneous disease causing itch (active eczema, urticaria or insect bites)
2. Active systemic disease that may induce itch (hepatic or renal disease).
3. Active psychiatric disease that could interfere with symptom assessment.
4. Treatment with drugs inducing itch.
5. Treatment with oral or topical preparations that could interfere with the itching sensation induced by patch test.
6. Treatment with systemic or topical corticosteroids, antihistaminics or calcineurin inhibitors.
7. Active skin disease in the back that may interfere with the assessment of response to topical application of allergen
8. Pregnancy or lactation
9. Subjects with contraindications specified in Summary of Product Characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Mean time to Itch Relief (TR) from the start of treatment, with methylprednisolone aceponate. | 5 days
  Time to Itch Relief is defined as the time needed to reach a 30% decrease of the maximum VAS (Visual Analogue Scale used for self-assessment of itch by the volunteers) recorded after the start of treatment.

SECONDARY OUTCOMES:
Erythema intensity by colorimetry. | 5 days
Eczema intensity by planimetric morphology (ICDRG scale) | 5 days
VAS versus time curve (time to reach VAS max from the start of treatment, AUC, dVAS/dT) | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Service, Hospital del Mar, Parc de Salut Mar, Barcelona, Barcelona, Spain